CLINICAL TRIAL: NCT04363931
Title: Investigation of the Effects of Kinesio Taping and Manual Therapy in Patients With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gokhan Yazici, Principal Investigator, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GaziU2020
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Bruxism
Keywords: Bruxism; Manual Therapy; Kinesio Taping; Physiotherapy
MeSH Terms: conditions — Bruxism | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Experimental): Manual Therapy is a widely used physiotherapy modality which is known to be effective in the management of musculoskeletal problems . Manual Therapy is a passive, therapeutic approach used to target a variety of anatomical structures with the intent to create beneficial changes in the amount of pain a patient experiences. Manual Therapy includes joint mobilization, manipulation, or treatment of the soft tissues and is widely used to break fibrous adhesions, restore normal range of motion, reduce local ischemia, stimulate synovial fluid production, and reduce pain .
  Interventions: Procedure: Manual Therapy
- Kinesio Taping (Experimental): Kinesio tape is a type of elastic therapeutic tape that was developed which is used in many different situations with various aims. Advocates of Kinesio Tape state that it may promote different therapeutic objectives such as; improved circulation and lymphatic drainage, pain inhibition, reduction of delayed onset of muscle soreness or improvement in performance and coordination .
  Interventions: Procedure: Kinesio Taping

INTERVENTIONS:
Procedure: Manual Therapy — Participants in this group received 4 weeks of manual therapy and massage of the masticatory muscles intra and extra orally together with massage of the cervical muscles. Massage and Manual Therapy brings about benefits by increasing local circulation and decreasing muscle tonus . Additionally, stretching exercises aiming to decrease pain and elongate shortened masticatory muscle fibers by autogenic inhibition of the masseter muscle were performed.
  Arms: Manual Therapy
Procedure: Kinesio Taping — Participants in this group had an application of Kinesio Taping on the masseter muscles. The material used for bruxism Kinesio Taping application was Kinesio Tex Gold Finger Prints (Kinesio Holding Corporation, Albuquerque, USA), a 100% cotton, latex-free, 5-cm wide, elastic tape. Kinesio Taping placement was chosen according to principles described by Kase et al. Tapes were cut 2.5 cm in width (cut in half vertically from 5 cm width). Two strips of Kinesio Tape were crossed over the masseter muscle area with 0-5% tension in maximum stretched epidermis position. Web-cut strips epidermis-dermis-fascia technique were used. Tape was applied bilaterally after every session of manual therapy.
  Arms: Kinesio Taping

SUMMARY:
Bruxism is defined as a repetitive jaw-muscle activity characterized by tooth grinding or clenching accompanied with wearing of the teeth, and jaw muscle discomfort in the absence of a medical disorder . Bruxism has two distinct circadian manifestations: it can be nocturnal or diurnal. Hypertrophy of the masseter muscle is an objective sign of bruxism. Additionally, fatigue or stiffness in the masticatory muscles, pain in the temporomandibular joint or headaches are subjective signs of bruxism. According to literature, 85% to 90% of the general population experience episodes of bruxism during their lives. Thus, finding an effective treatment method for bruxism is crucial.The aim of this study is to investigate the effects of two different physiotherapy approaches on the masseter muscle thickness and stiffness in patients with Bruxism.

DETAILED DESCRIPTION:
There is no certain treatment for Bruxism. However, the most recent recommendation is to follow the Multiple-P approach prior to medical drug regimens and invasive procedures. Different methods used in the conservative management of Bruxism are known as the "multiple-P" approach, which consists of; physiotherapy, plates, pep talk, pills and psychology . Physiotherapy generally focuses on two objectives: decreasing the adverse effects of bruxism to the masticatory muscles and increasing self-awareness regarding this habit. These studies involve different intervention such as massage of the masticatory and cervical muscles, electrotherapy, therapeutic exercises, taping interventions or relaxation therapies . However, literature regarding which physiotherapy intervention is the most effective in bruxism is not clear. Therefore patients in this study were randomly divided into one of two groups; manual therapy or kinesio taping. All patients were assessed at baseline, received 4 weeks of treatment and were assessed following the 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A Bruxism Diagnosis according to the criteria of the international classification for sleep disorders
* Self-report of awake bruxism

Exclusion Criteria:

* Having more than 2 missing teeth
* The presence of removable partial dentures
* Having neurological, psychiatric or motor disorders
* Having any ongoing dental or physical therapy
* Active cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold of Masseter Muscle | Change from Baseline Pain Pressure Threshold of Masseter Muscle at 4 weeks
  Pain Pressure Threshold was determined using a digital algometer (Lafayette Manual Muscle Test System™, Model 01163, Lafayette Instrument Company, Indiana, USA) which consists of a padded disc attached to a microprocessor control unit that measures peak force (Newton). The Pain Pressure Threshold of the masseter muscle was assessed via the algometer. During Pain Pressure Threshold assessment, the researcher positioned the algometer on the trigger points of the respective muscle and increase the amount of pressure applied until the participant verbally informed the researcher when the sensation of pressure became pain. The applied pressure was read from the digital screen after each assessment.
Pain Pressure Threshold of Trapezius Muscle | Change from Baseline Pain Pressure Threshold of Trapezius Muscle at 4 weeks
  Pain Pressure Threshold was determined using a digital algometer (Lafayette Manual Muscle Test System™, Model 01163, Lafayette Instrument Company, Indiana, USA) which consists of a padded disc attached to a microprocessor control unit that measures peak force (Newton). The Pain Pressure Threshold of the trapezius muscle was assessed via the algometer. During Pain Pressure Threshold assessment, the researcher positioned the algometer on the trigger points of the respective muscle and increase the amount of pressure applied until the participant verbally informed the researcher when the sensation of pressure became pain. The applied pressure was read from the digital screen after each assessment.
Pain Pressure Threshold of Temporalis Muscle | Change from Baseline Pain Pressure Threshold of Temporalis Muscle at 4 weeks
  Pain Pressure Threshold was determined using a digital algometer (Lafayette Manual Muscle Test System™, Model 01163, Lafayette Instrument Company, Indiana, USA) which consists of a padded disc attached to a microprocessor control unit that measures peak force (Newton). The Pain Pressure Threshold of the temporalis muscle was assessed via the algometer. During Pain Pressure Threshold assessment, the researcher positioned the algometer on the trigger points of the respective muscle and increase the amount of pressure applied until the participant verbally informed the researcher when the sensation of pressure became pain. The applied pressure was read from the digital screen after each assessment.

SECONDARY OUTCOMES:
Sleep Quality | Change from Baseline Sleep Quality at 4 weeks
  The Pittsburgh Sleep Quality Index is an index widely used to measure sleep quality. The Pittsburgh Sleep Quality Index is a self-reported questionnaire that includes 19 questions that when scored, are separated into seven domains. The seven domains are; perceived sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medications; and daytime dysfunction. Each domain is scored from 0-3 and a total score ranging from 0-21 can be obtained. A total score of; 0-4 indicates a good sleep quality, 5-10 indicates poor sleep quality and scores above 10 indicate a possible sleep disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yazici, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers